CLINICAL TRIAL: NCT01128595
Title: A Randomised, Double-blind, Placebo-controlled, Four-way Crossover, Repeat Dose Study Comparing the Effect of Inhaled Fluticasone Furoate/GW642444M Combination, GW642444M and Fluticasone Furoate on the Allergen-induced Asthmatic Response in Subjects With Mild Asthma
Brief Title: Randomised Study Comparing the Effects of Inhaled FF/GW642444M Combination, FF and GW642444M on an Allergen Induced Asthmatic Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113126
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: allergen challenge; early asthmatic response; mild asthma; late asthmatic response
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ICS (Active Comparator)
  Interventions: Drug: Fluticasone Furoate
- ICS/LABA (Active Comparator)
  Interventions: Drug: FF/GW642444M
- LABA (Active Comparator)
  Interventions: Drug: GW642444M
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FF/GW642444M
  Arms: ICS/LABA
Drug: GW642444M
  Arms: LABA
Drug: Fluticasone Furoate
  Arms: ICS
Drug: Placebo
  Arms: Placebo

SUMMARY:
We propose to use an inhaled allergen challenge model to explore the individual contributions of the components of a novel long-acting beta agonist/ inhaled corticosteroid combination product and its components on protection from allergic triggers in asthma

DETAILED DESCRIPTION:
Asthma is an increasingly common disease and is essentially caused by an allergic type of reaction of the immune system. Airways of the lungs become inflamed and narrow as a result of a reaction to triggers like chemicals (house-hold cleaning products, pollution) and allergens (house dust mite and cat or dog fur). The airways become blocked, causing shortness of breath and wheezing. The purpose of this study is to find out more information about how effective the study drugs are at protecting the lungs against allergic triggers of asthma. There are three study drugs being investigated in this study: fluticasone furoate on its own, GW642444M on its own and a combination of fluticasone furoate (FF) and GW642444M.

FF is a corticosteroid that is being developed by for the treatment of asthma. A nasal spray formulation of FF has been approved for marketing in the USA, Europe and Japan for the treatment of hayfever (rhinitis) but the dry powder formulation used in this study is not yet approved.

GW642444M is a long-acting beta2-agonist being developed by GSK for the treatment of chronic obstructive pulmonary disease (COPD). It works by acting on cells in the lungs, causing some of the muscles around the lungs to relax and open up better (bronchodilation), making breathing easier. The combination of FF/GW642444M is being developed as a once-daily treatment for both asthma and COPD.

Study treatment will be taken for 21 days in each period (4 treatment periods: FF alone, GW642444M alone, FF/GW64244M combination and placebo) and each subject will receive all treatments. On D21 subjects will undergo an allergen challenge, followed by a methacholine challenge on D22. The washout between treatment periods will be 21-35 days.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index within the range 18.5-35.0 kilograms/metre2 (kg/m2).

* Females of non-child bearing potential.
* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta -agonist therapy by inhalation
* Pre-bronchodilator FEV1 >70% of predicted at screening
* Subjects who are current non-smokers
* Methacholine challenge PC20 < 8 mg/mL at screening
* Screening allergen challenge demonstrates that the subject experiences an early asthmatic response

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities

  * Subject is hypertensive at screening
  * Respiratory tract infection and/or exacerbation of asthma within 4 weeks prior to the first dose of study medication.
  * History of life-threatening asthma
  * Symptomatic with hay fever at screening or predicted to have symptomatic hayfever
  * Unable to abstain from short acting beta agonists
  * Unable to abstain from antihistamines
  * Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDs), anti-depressant drugs, anti-asthma anti-rhinitis or hay fever medication
  * The subject has participated in a study with a new molecular entity during the previous 3 months or has participated in 4 or more clinical studies in the previous 12 months
  * undergoing allergen desensitisation therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Randwick, New South Wales, Australia
- GSK Investigational Site, Wellington, New Zealand
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113126 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113126 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113126 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113126 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113126 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113126 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113126 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting all of the inclusion criteria and none of the exclusion criteria during the Screening Visit, conducted 14-42 days prior to the first dose of study medication, entered a 14-day Run-in Period. Participants were then randomized to 4 Treatment Periods, each lasting 21 days and separated by a nominal washout period of 21-35 days.
Groups:
- Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg: Participants received Vilanterol (VI) 25 micrograms (µg), placebo, fluticasone furoate (FF) 100 µg, and FF/VI 100/25 µg in Treatment Periods 1, 2, 3, and 4, respectively. Participants received all treatments once a day (OD) for 21 days from a Dry Powder Inhaler (DPI). The four treatment periods were separated by a washout period of 21 to 35 days.
- Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg: Participants received FF/VI 100/25 µg, FF 100 µg, placebo, and VI 25 µg in Treatment Periods 1, 2, 3, and 4, respectively. Participants received all treatments once a day (OD) for 21 days from a Dry Powder Inhaler (DPI). The four treatment periods were separated by a washout period of 21 to 35 days.
- Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg: Participants received placebo, FF/VI 100/25 µg, VI 25 µg, and FF 100 µg in Treatment Periods 1, 2, 3, and 4, respectively. Participants received all treatments once a day (OD) for 21 days from a Dry Powder Inhaler (DPI). The four treatment periods were separated by a washout period of 21 to 35 days.
- Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo: Participants received FF 100 µg, VI 25 µg, FF/VI 100/25 µg, and placebo in Treatment Periods 1, 2, 3, and 4, respectively. Participants received all treatments once a day (OD) for 21 days from a Dry Powder Inhaler (DPI). The four treatment periods were separated by a washout period of 21 to 35 days.
Period: Treatment Period 1
Arm/Group | Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg | Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg | Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo
Started | 7 | 6 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg | Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg | Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo
Started | 7 | 6 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg | Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg | Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo
Started | 7 | 6 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg | Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg | Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo
Started | 7 | 6 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg | Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg | Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo
Started | 7 | 6 | 7 | 7
Completed | 7 | 5 | 7 | 7
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Washout Period 3
Arm/Group | Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg | Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg | Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo
Started | 7 | 5 | 7 | 7
Completed | 7 | 5 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Sequence 1: VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg | Sequence 2: FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg | Sequence 3: Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg | Sequence 4: FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo
Started | 7 | 5 | 7 | 7
Completed | 7 | 5 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo, FF/VI 100/25 µg OD, FF 100 µg OD, VI 25 µg: All participants received one of the following four treatments in one of four treatment periods once daily (OD) from the Dry Powder Inhaler (DPI) for 21 days: Placebo; Fluticasone Furoate /Vilanterol (FF/VI) 100/25 microgram (µg) dry inhalation powder; Fluticasone Furoate (FF) 100 µg dry inhalation powder; and Vilanterol (VI) 25 µg dry inhalation powder. Participants were randomized to receive treatment in one of the four following sequences: (1) VI 25 µg, Placebo, FF 100 µg, FF/VI 100/25 µg; (2) FF/VI 100/25 µg, FF 100 µg, Placebo, VI 25 µg; (3) Placebo, FF/VI 100/25 µg, VI 25 µg, FF 100 µg; (4) FF 100 µg, VI 25 µg, FF/VI 100/25 µg, Placebo. The four treatment periods were separated by a washout period of 21 to 35 days.
Arm/Group | Placebo, FF/VI 100/25 µg OD, FF 100 µg OD, VI 25 µg
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.8 (7.46)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian/European Heritage | 25
  East Asian Heritage | 1
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Late Asthmatic Response (LAR): Absolute Change From Saline in Minimum FEV1 Between 4-10 Hours (Hrs) Following the 1-hr Post-treatment Allergen Challenge on Day 21 of Each Treatment Period
Description: Forced expiratory volume in one second (FEV1) is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen (administered by inhalation) 1 hr after dosing on Day 21. Minimum FEV1 over 4-10 hours post-allergen challenge (minimum LAR) is the minimum value of all of the post-saline time points between 4 and 10 hrs post-allergen challenge, inclusive of the 4 hr and 10 hr timepoints (i.e., minimum over 4 hrs, 4.5 hrs, 5 hrs, 5.5 hrs, 6 hrs, 6.5 hrs, 7 hrs, 7.5 hrs, 8 hrs, 8.5 hrs, 9 hrs, 9.5 hrs, and 10 hrs). Absolute change from saline in minimum FEV1 was calculated as the minimum FEV1 minus the saline FEV1 value. After inhalation of saline, 3 single measurements of FEV1 were recorded; the maximum FEV1 value was taken as the saline value. Least squares means were obtained by adjusting for period and participant and period Baselines.
Time Frame: Day 21 of each treatment period (up to Study Day 197)
Population: Efficacy Population: all participants who received at least one dose of study medication, had a post-dose FEV1 assessment, and who were not major protocol violators. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- FF/VI 100/25 µg OD: Participants received FF/VI 100/25 µg OD from the DPI for 21 days during one of the four treatment periods. Each treatment period was followed by a washout period of 21-35 days.
- FF 100 µg OD: Participants received FF 100 µg OD from the DPI for 21 days during one of the four treatment periods. Each treatment period was followed by a washout period of 21-35 days.
- VI 25 µg OD: Participants received VI 25 µg OD from the DPI for 21 days during one of the four treatment periods. Each treatment period was followed by a washout period of 21-35 days.
Arm/Group | Placebo | FF/VI 100/25 µg OD | FF 100 µg OD | VI 25 µg OD
Number analyzed (Participants) | 20 | 26 | 27 | 22
Liters | -0.731 [-0.878 to -0.584] | -0.216 [-0.343 to -0.088] | -0.188 [-0.315 to -0.061] | -0.536 [-0.676 to -0.396]
Statistical Analysis 1: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.515, 95% CI 2-sided [0.330 to 0.701]
Statistical Analysis 2: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.543, 95% CI 2-sided [0.355 to 0.730]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.195, 95% CI 2-sided [0.001 to 0.388]
Statistical Analysis 4: Comparison: FF/VI 100/25 µg OD vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.027, 95% CI 2-sided [-0.198 to 0.143]
Statistical Analysis 5: Comparison: FF/VI 100/25 µg OD vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.320, 95% CI 2-sided [0.140 to 0.501]

2. Secondary Outcome: Maximum Percent Change From Saline in FEV1 Between 0-2 Hrs, Following the 1-hr Post-treatment Allergen Challenge on Day 21 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 1 hr after dosing on Day 21. FEV1 was measured 0 minutes (min), 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 hr, 1.5 hrs, and 2 hrs post-allergen challenge on Day 21. Maximum percent change was calculated as the minimum FEV1 minus the saline FEV1 value divided by the saline FEV1 multiplied by 100. After inhalation of saline, 3 single measurements of FEV1 were recorded; the maximum FEV1 value was taken as the saline FEV1 value.
Time Frame: Day 21 of each treatment period (up to Study Day 197)
Population: Efficacy Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: percent change
Groups:
- Placebo: Participants received placebo OD from the DPI for 21 days during one of the four treatment periods. Each treatment period was followed by a washout period of 21-35 days.
Arm/Group | Placebo | FF/VI 100/25 µg OD | FF 100 µg OD | VI 25 µg OD
Number analyzed (Participants) | 22 | 27 | 27 | 22
percent change | -26.13 [-58.9 to -5.4] | -10.43 [-58.9 to -2.1] | -16.14 [-64.9 to -4.0] | -18.35 [-59.3 to -4.4]

3. Secondary Outcome: Provocative Concentration of Methacholine Estimated to Result in a 20% Reduction in FEV1 (PC20) on Day 22 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants inhaled doubling increments of methacholine until a >=20% fall in FEV1 from the saline value was achieved. After inhalation of saline, 3 measurements of FEV1 were recorded; the maximum FEV1 value was taken as the saline value.
Time Frame: Day 22 of each treatment period (up to Study Day 198)
Population: Efficacy Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: milligrams per milliliter
Arm/Group | Placebo | FF/VI 100/25 µg OD | FF 100 µg OD | VI 25 µg OD
Number analyzed (Participants) | 23 | 27 | 25 | 24
milligrams per milliliter | 1.046 (3.3191) | 2.500 (3.7363) | 2.492 (5.3371) | 0.387 (0.5311)

4. Primary Outcome: LAR: Absolute Change From Saline in Weighted Mean (WM) FEV1 Between 4-10 Hrs Following the 1-hr Post-treatment Allergen Challenge on Day 21 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 1 hour after dosing on Day 21. LAR FEV1 was measured 4 hrs, 4.5 hrs, 5 hrs, 5.5 hrs, 6 hrs, 6.5 hrs, 7 hrs, 7.5 hrs, 8 hrs, 8.5 hrs, 9 hrs, 9.5 hrs, and 10 hrs post-allergen challenge on Day 21. Absolute change from saline in WM FEV1 was calculated as the area under the curve divided by the relevant time interval and subtracting the saline FEV1 value. After inhalation of saline, 3 single measurements of FEV1 were recorded; the maximum FEV1 value was taken as the saline value. Least squares means were obtained by adjusting for period and participant and period Baselines.
Time Frame: Day 21 of each treatment period (up to Study Day 197)
Population: Efficacy Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FF/VI 100/25 µg OD | FF 100 µg OD | VI 25 µg OD
Number analyzed (Participants) | 20 | 26 | 27 | 22
Liters | -0.466 [-0.589 to -0.343] | 0.018 [-0.089 to 0.125] | 0.018 [-0.089 to 0.124] | -0.298 [-0.415 to -0.181]
Statistical Analysis 1: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.484, 95% CI 2-sided [0.332 to 0.636]
Statistical Analysis 2: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.484, 95% CI 2-sided [0.330 to 0.638]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.168, 95% CI 2-sided [0.009 to 0.327]
Statistical Analysis 4: Comparison: FF/VI 100/25 µg OD vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.000, 95% CI 2-sided [-0.140 to 0.140]
Statistical Analysis 5: Comparison: FF/VI 100/25 µg OD vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.316, 95% CI 2-sided [0.168 to 0.464]

5. Primary Outcome: Early Asthmatic Response (EAR): Absolute Change From Saline in Minimum FEV1 Between 0-2 Hrs Following the 1-hr Post-treatment Allergen Challenge on Day 21 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 1 hr after dosing on Day 21. Minimum FEV1 over 0-2 hrs post-allergen challenge (Minimum EAR) is the minimum value of all of the post-allergen challenge timepoints up to and including 2 hours post-allergen challenge (i.e., minimum over 5 minutes (min), 10 min, 15 min, 20 min, 30 min, 45 min and 1 hr, 1.5 hrs, and 2 hrs. Absolute change from saline in minimum FEV1 was calculated as the minimum FEV1 minus the saline FEV1 value. After inhalation of saline, 3 single measurements of FEV1 were recorded; the maximum FEV1 value was taken as the saline value. Least squares means were obtained by adjusting for period and participant and period Baselines.
Time Frame: Day 21 of each treatment period (up to Study Day 197)
Population: Efficacy Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FF/VI 100/25 µg OD | FF 100 µg OD | VI 25 µg OD
Number analyzed (Participants) | 22 | 27 | 27 | 22
Liters | -1.091 [-1.344 to -0.837] | -0.614 [-0.858 to -0.370] | -0.826 [-1.070 to -0.581] | -0.955 [-1.209 to -0.702]
Statistical Analysis 1: Comparison: FF/VI 100/25 µg OD vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.212, 95% CI 2-sided [0.031 to 0.393]
Statistical Analysis 2: Comparison: FF/VI 100/25 µg OD vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.341, 95% CI 2-sided [0.147 to 0.536]
Statistical Analysis 3: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.477, 95% CI 2-sided [0.282 to 0.672]
Statistical Analysis 4: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.265, 95% CI 2-sided [0.066 to 0.463]
Statistical Analysis 5: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.135, 95% CI 2-sided [-0.072 to 0.343]

6. Primary Outcome: EAR: Absolute Change From Saline in Weighted Mean FEV1 Between 0-2 Hrs Following the 1-hr Post-treatment Allergen Challenge on Day 21 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 1 hr after dosing on Day 21. The EAR FEV1 was measured 0 minutes (min), 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 hr, 1.5 hrs, and 2 hrs post-allergen challenge on Day 21. Least squares means were obtained by adjusting for period and participant and period Baselines. Absolute change from saline in WM FEV1 was calculated as the area under the curve divided by the relevant time interval and subtracting the saline FEV1 value. After inhalation of saline, 3 single measurements of FEV1 were recorded; the maximum FEV1 value was taken as the saline value.
Time Frame: Day 21 of each treatment period (up to Study Day 197)
Population: Efficacy Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FF/VI 100/25 µg OD | FF 100 µg OD | VI 25 µg OD
Number analyzed (Participants) | 22 | 27 | 27 | 22
Liters | -0.560 [-0.745 to -0.374] | -0.297 [-0.476 to -0.118] | -0.386 [-0.565 to -0.207] | -0.533 [-0.718 to -0.348]
Statistical Analysis 1: Comparison: FF/VI 100/25 µg OD vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.089, 95% CI 2-sided [-0.037 to 0.215]
Statistical Analysis 2: Comparison: FF/VI 100/25 µg OD vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.236, 95% CI 2-sided [0.101 to 0.371]
Statistical Analysis 3: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.263, 95% CI 2-sided [0.127 to 0.398]
Statistical Analysis 4: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [0.036 to 0.312]
Statistical Analysis 5: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.118 to 0.171]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the fourth treatment period (up to Day 210).
Description: SAEs and non-serious AEs were reported for members of the All Participants Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | FF/VI 100/25 µg OD | FF 100 µg OD | VI 25 µg OD
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 19/27 | 20/27 | 19/27 | 22/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | FF/VI 100/25 µg OD (N=27) | FF 100 µg OD (N=27) | VI 25 µg OD (N=26)
Headache (Nervous system disorders) | 11 | 15 | 15 | 13
Nasopharyngitis (Infections and infestations) | 2 | 3 | 2 | 5
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Eczema infected (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Eye penetration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 3 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.